CLINICAL TRIAL: NCT06329492
Title: Autologous Alpha-2 Macroglobulin Rich Plasma (A2MRP), Safety and Efficacy in Symptomatic Moderate Knee Osteoarthritis: A Pilot Study
Brief Title: Autologous Alpha-2 Macroglobulin Rich Plasma, Safety and Efficacy in Symptomatic Moderate Knee Osteoarthritis
Acronym: A2MRP
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Brennan J. Boettcher, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 23-007937
Record Dates: First submitted 2024-02-27; First posted 2024-03-26 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Osteoarthritis; OA; Knee Osteoarthritis
Keywords: regenerative med
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee

STUDY DESIGN:
Intervention Model Description: Single group cohort of 20 subjects
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Autologous Alpha-2 Macroglobulin Rich Plasma (A2MRP) (Experimental): Autologous Alpha-2 Macroglobulin Rich Plasma (A2MRP) is produced by filtering Platelet Poor Plasma (PPP), a Platelet Rich Plasma byproduct, through a hemoconcentrator filter. (PPP) is frequently used in clinical practice to increase volume of PRP or Bone Marror Aspirate Concentrate (BMAC) injectate, and it is occasionally injected in isolation for some indication
  Interventions: Biological: Autologous Alpha-2 Macroglobulin Rich Plasma (A2MRP)

INTERVENTIONS:
Biological: Autologous Alpha-2 Macroglobulin Rich Plasma (A2MRP) — Your blood will be processed into Autologous Alpha-2 Macroglobulin Rich Plasma (A2MRP) A2MRP in the procedure room with you while you wait. This will take approximately 30 minutes. When this is complete, an ultrasound will be done of your knee to determine the best location for injection into the knee joint. You will undergo an ultrasound guided injection, and the needle guided into the knee joint, and the Autologous Alpha-2 Macroglobulin Rich Plasma (A2MRP) A2MRP will be injected into the joint space. If there is excessive fluid in your knee, this may be drained before the injection is performed. The needle will be removed, and a band aid will be placed over the injection site.

SUMMARY:
The purpose of this study is to determine the effectiveness and safety of autologous alpha-2 macroglobulin rich plasma (A2MRP) injections in the treatment of knee osteoarthritis (OA).

DETAILED DESCRIPTION:
The overall objective of this study is to test and quantify A2MRP and prepare for a larger randomized clinical trial assessing the efficacy of A2MRP injections in primary and post traumatic knee osteoarthritis (OA) with respect to clinical outcomes and disease progression. The study will also assess safety of A2MRP intraarticular injection in patients with symptomatic knee OA. Patients with symptomatic mild to moderate knee OA (KL 2-3) will be candidates for this study. Baseline data will include physical examination of the knee, clinical assessment of knee pain and function using validated patient reported outcome measures (PROMs), and radiologic exam of the knee will be obtained. All injections will be performed using ultrasound guidance and all patients will followed-up at week 1 week post-injection for acute adverse events (AEs). Each subject will be clinically followed-up for study endpoints using a predetermined protocol. PROs will be collected during the study period pre-procedure, and at 1, 2, and 6 weeks, 3-, 6-, 9- and 12-months post-procedure (Specific PRO's and timepoints noted in sections 6.2-6.7). Subjects will also be asked questions regarding satisfaction with the treatment and whether they would recommend the treatment

ELIGIBILITY:
Inclusion Criteria:

1. Male or females,18-65 years of age
2. Chronic (> 3 months), unilaterally symptomatic, primary knee OA.
3. Painful knee OA in one or more knee compartments grade 2-3 radiologic severity based upon the Kellgren-Lawrence grading scale, without evidence of advanced (bone on bone, as determined by study investigators) OA in the patellofemoral compartment or on Posterior Anterior (PA) flexion views
4. Cognitive ability to give informed consent
5. Speak fluent English
6. Worst knee pain greater than 4 on a 0-10 pain scale (0 = no pain, 10 = worst pain imaginable)
7. Previous 6 week or longer trial of one of the following conservative treatments: activity modification, weight loss, physical therapy, anti-inflammatory medications/acetaminophen or injection therapy (e.g., cortisone)
8. Fully understanding of the requirements of the study and willingness to comply with the treatment plan, including blood draw, laboratory tests, diagnostic imaging, and follow-up visits and assessments
9. Can provide written informed consent and complete HIPAA documentation after the nature of the study is fully explained and prior to any study-related procedure.

Exclusion Criteria:

1. Pregnant or nursing, or planning on becoming pregnant during the study period
2. Congenital or acquired malformation of the target knee resulting in significant deformity or leading to problems with the study treatment or analysis of the results
3. Significant valgus or varus malalignment as determined by investigator
4. Injections of any kind into the target knee:

   * Corticosteroid injections within 3 months prior to study enrollment
   * Hyaluronic acid injections within 6 months prior to study enrollment
   * PRP injection within the year prior to study enrollment
   * History of BMAC, Micro-Fragmented Adipose Tissue (MFAT), or perinatal product injection at any point
5. History of intra-articular infection in the target knee
6. History of superficial infection in the target knee within 6 months of study enrollment, or evidence of current superficial infection affecting the target knee
7. Body mass index (BMI) < 35 kg/m2
8. Inability to stop non-steroidal anti-inflammatory medications for 1 week before through 2 weeks after the procedure date
9. On chronic, immunosuppressive transplant therapy or having a chronic, immunosuppressive state, including use of systemic steroids/corticosteroids
10. Current tobacco product use, including nicotine patch or other nicotine products
11. Clinically significant rheumatological or inflammatory disease or chondrocalcinosis/ calcium pyrophosphate disease (CPPD), hemochromatosis, inflammatory arthritis, arthropathy of the knee associated with juxta-articular Paget's disease of the femur or tibia, ochronosis, hemophilic arthropathy, systemic sclerosis, system lupus erythematosus, and Ehlers-Danlos Syndrome, infectious arthritis, Charcot's knee joint, villonodular synovitis, and synovial chondromatosis
12. Surgery in the target knee within the last 12 months, or planned surgery in the target knee in next 12 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2024-01-09 (Actual); Primary Completion 2026-01-28 (Actual); Study Completion 2026-02-06 (Actual)

PRIMARY OUTCOMES:
Adverse Events | 1 year
  The number of Adverse Events reported

SECONDARY OUTCOMES:
Visual Analog Scale (VAS) for Pain | 1 year
  The VAS is a 11-item questionnaire assessing pain. Using a scale of 0 = no pain to 10 = worst pain. Total scores range from 0 - 110, lower scores indicating lower pain and higher scores indicating greater pain.
Patient-Reported Outcomes Measurement Information System (PROMIS)-Computer adaptive test (CAT): Pain interference | 1 year
  The PROMIS-CAT: Pain interference is a 40-item questionnaire assessing pain. Using a scale of 1 = not at all to 5 = very much. Total scores range from 40-200, lower scores indicating lower pain and higher scores indicating greater pain.
Patient-Reported Outcomes Measurement Information System (PROMIS)-Computer adaptive test (CAT): Physical function | 1 year
  The PROMIS-CAT: Physical function is a 165-item questionnaire assessing physical function. Using a scale of 1 = unable to do to 5 = without any difficulty. Total scores range from 165-825, lower scores indicating less physical function and higher scores indicating greater physical function.
Knee Injury and Osteoarthritis Outcome Score (KOOS): | 1 year
  KOOS is a commonly used questionnaire which focuses on how patients are affected by knee problems in five areas: knee pain, stiffness, daily activity, sport and recreation, and quality of life. Results are scored 0-100. 0 = extreme knee problems, 100 = no knee problems
Procedure Recommendation | 1 year
  The number of subjects to answer "yes" to the question "Would you recommend this procedure to someone with a similar condition as your own?"

CONTACTS AND LOCATIONS:
Overall Officials: Brennan Boettcher, D.O, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Mayo Clinic Clinical Trials — https://www.mayo.edu/research/clinical-trials/list-studies